CLINICAL TRIAL: NCT00098072
Title: Endothelial Cell Dysfunction in Pulmonary Arterial Hypertension: Biomarkers, Mechanisms of Disease and Novel Therapeutic Targets
Brief Title: Endothelial Cell Dysfunction in Pulmonary Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 050041; 05-CC-0041
Record Dates: First submitted 2004-12-02; First posted 2004-12-03 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-09

CONDITIONS: Secondary Pulmonary Arterial Hypertension
Keywords: Cytometry; Genes; Hypertension; Lung; Proteomics; Primary Pulmonary Hypertenion; PPH; Healthy Volunteers; HV
MeSH Terms: conditions — Hypertension | interventions — Cardiac Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): Pilot
  Interventions: Procedure: Heart Catheterization

INTERVENTIONS:
Procedure: Heart Catheterization — Heart Catheterization and collection of samples

SUMMARY:
This study will examine and test healthy volunteers and patients with pulmonary hypertension to try to learn more about the disease and find better ways to detect, treat, and, if possible, slow progression. Pulmonary hypertension is a rare blood vessel disorder of the lung in which the pressure in the pulmonary artery (the blood vessel that leads from the heart to the lungs) rises above normal levels and may become life-threatening.

Normal volunteers and patients with pulmonary hypertension 18 years of age and older may be eligible for this study. All candidates are screened with a review of their medical records. Normal volunteers also have a medical history, electrocardiogram, echocardiogram (heart ultrasound), and pulmonary function test, in which the subject breathes in and out of a tube that measures lung volume, mechanics and function.

All participants undergo the following tests and procedures:

* Echocardiogram to measure heart function and blood pressure in the lungs. A small probe held against the chest uses sound waves to obtain pictures of the heart.
* Magnetic resonance imaging (MRI) to evaluate the heart's pumping action. Subjects lie on a stretcher that slides into a long, tube-shaped scanner. The machine uses a magnetic field and radio waves to obtain images of the heart.
* 6-minute walk to measure how far the subject can walk in 6 minutes. Subjects walk around the hospital for 6 minutes at a comfortable pace.
* Exercise testing to measure the ability to exercise and the subject's oxygen levels during exercise. Subjects exercise on a bike or treadmill while the oxygen and carbon dioxide they breathe are measured using a small device placed in the mouth.
* Right heart catheterization to measure pressure in the heart and lungs. A small catheter (plastic tube) is placed in an arm vein. A longer catheter called a central line is placed in a deeper vein in the neck or just below the neck, or in the leg or arm. A long, thin catheter that measures blood pressure directly is then inserted into the vein and advanced through the chambers of the heart into the lung artery to measure all the pressures in the heart and obtain blood samples.
* Genetic and protein studies. DNA, RNA, and proteins from blood samples are studied for genes and proteins that might predict the development or progression of pulmonary hypertension.

In addition to the above, patients whose pulmonary hypertension was caused by a blood vessel injury undergo the tests described below. The right heart catheter inserted for the catheterization procedure remains in place to obtain measurements of the effects of nitric oxide and nitrite in the following procedures:

* Inhalation of nitric oxide (a gas naturally produced by cells lining arteries) at 30-minute intervals to examine its effect on lung and heart pressures.
* Inhalation of aerosolized nitrite at 5-minute intervals to measure its effects on lung and heart pressures.
* Inhalation of nitric oxide for up to 24 hours to obtain multiple measurements of its effect on lung and heart pressures.
* Blood draws for laboratory tests.

In patients whose pulmonary hypertension was caused by a blood vessel injury, we also plan to follow response to standard therapy. After the initiation of standard therapy, we will restudy the same parameters (excluding NO and sodium nitrite studies) in these patients at approximately 4 months, and yearly for 5 years

...

DETAILED DESCRIPTION:
Introduction: Primary pulmonary hypertension, now known as idiopathic pulmonary arterial hypertension (IPAH), a subgroup of pulmonary arterial hypertension (PAH), is a rare disorder characterized by severe morbidity and high mortality rates. There are no routine screening tests or validated markers of disease activity in IPAH, or the broader group of PAH. Therefore, patients usually present at advanced stages of disease. The pathogenesis of IPAH and other forms of PAH remain unclear. Prior theories stressed a "one-hit" hypothesis. Current thinking focuses on a "two-hit" hypothesis: 1) genetic susceptibility, and 2) a triggering stimulus that initiates pulmonary vascular injury, resulting in endothelial cell (EC) dysfunction and the mobilization of endothelial progenitor cells (EPC). Loss of function mutations in the bone morphogenetic protein receptor 2 (BMPR2) gene, has been implicated in the pathogenesis of IPAH. EC dysfunction in IPAH has been associated with decreases in both endothelial nitric oxide synthase (eNOS) expression and nitric oxide (NO) production. Peripheral blood mononuclear cells (PBMCs) interact with an altered endothelial cell surface, which may also be important in the disease process.

Objectives: We plan to define a subset of differentially regulated biomarkers in IPAH and PAH that may lead to earlier diagnosis and better methods for measuring responses to therapy. Specifically, we hope to identify biomarkers of IPAH and other forms of PAH that is suggestive of NO therapeutic response and which may be useful in titrating NO therapy. We also hope to identify novel targets for the development of new therapeutic strategies.

Methods: This study will consist of a pilot study and a primary study. The pilot study will enroll up to 30 patients and 30 controls in order to obtain completed studies on 10 normal subjects and 10 patients with PAH. The goal of the pilot study is to determine the best technique for circulating endothelial cell (CEC) and PBMC identification, quantification, and isolation and EPC identification and quantification. The subjects in the pilot phase undergo right heart catheterization to obtain hemodynamics and pulmonary artery blood. Pulmonary artery and peripheral blood will be used for EPC quantification and CEC and PBMC isolation. CECs and PBMCs will be studied in depth using high density oligonucleotide microarrays. In addition, plasma obtained from PAH patients and healthy volunteers will be applied in vitro to various cell populations suspected to be central to disease pathogenesis including but not limited to ECs, circulating mononuclear cells, cardiac myocytes and/or vascular smooth muscle cells. Phenotypic alterations induced by plasma exposure will be assessed using in vitro assays.

The primary study will recruit the following subject groups: 1) patients with IPAH and other forms of PAH (vascular injury-induced pulmonary hypertension) who currently are on no therapy, less than or equal to 6 months of IV therapy, or less than or equal to one year of oral therapy, 2) patients with pulmonary hypertension (PH) ascribed to a nonvascular injury process and 3) normal individuals. The following baseline studies will be performed in all groups: 1) noninvasive assessment of right ventricular (RV) function by echocardiogram and magnetic resonance imaging (MRI), 2) determination of exercise capacity by cardiopulmonary stress test and six minute walk, 3) measurement of hemodynamic parameters by right heart catheterization and 4) characterization of disease phenotype by cell surface markers, oligonucleotide microarrays, and proteomics using peripheral and pulmonary arterial blood. EPCs will be quantitated and CECs and PBMCs will be isolated and analyzed by flow cytometry for expression of cell surface markers involved in coagulation, adhesion, and angiogenesis, as these are important processes in IPAH and PAH. Furthermore, ECs (identified by positive and negative selection and isolated by cell sorting) and PBMCs will be studied in depth using high density oligonucleotide microarrays to more fully characterize their transcriptome.

A major impediment to the widespread use of chronic home based inhaled NO are related to its delivery system and duration of effects. In PAH patients we plan to study a novel NO delivery system (INO pulse delivery device). Patients with PAH will be given inhaled NO (20 and 40 ppm) and then placed on inhaled NO using the INO pulse delivery device for 24 hours. Hemodynamics will be obtained serially with each dose and upon completion of 24 hours of therapy, pulmonary artery and peripheral blood will be drawn and reexamined by flow cytometry, microarrays, and proteomics.

We also plan to follow response to standard therapy (as determined by the referring physician). After the initial day 0 studies, we will restudy the same parameters (excluding NO studies) in patients with PAH at approximately 4 months, and yearly for 5 years after therapeutic intervention.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Pilot: The pilot study will enroll two groups of individuals: 1) patients who have either IPAH or a secondary form known to have similar histopathology (PAH), and 2) age, gender, and race matched control subjects for each patient.

Main: The main study will enroll three groups of individuals: 1) patients who have either IPAH or a secondary form known to have similar histopathology (PAH), 2) patients with PH ascribed to a nonvascular injury process, and 3) age, gender, and race matched control subjects for each PAH patient. Subjects must be at least 18 years of age and must be able to provide informed, written consent for participation in this study. There is no exclusion based on race or gender.

INCLUSION CRITERIA FOR PULMONARY ARTERIAL HYPERTENSION PATIENTS:

The inclusion criteria for this study are as follows:

1. Patients diagnosed with IPAH
2. Patients diagnosed with secondary pulmonary hypertension known to have histopathology similar to the primary form or PAH. Clinical conditions causing pulmonary hypertension with histopathology similar to the primary form are listed below.

   i. Eisenmenger Syndrome

   ii. Collagen vascular disease

   iii. Liver disease with portal hypertension

   iv. Toxin induced injury (anorexic agents, rapeseed oil)

   v. HIV disease

   vi. Sickle cell disease

   EXCLUSION CRITERIA FOR PATIENTS WITH PULMONARY ARTERIAL HYPERTENSION:

<!-- -->

1. Pregnant women (all women of childbearing age will be required to have a screening urine or blood pregnancy test)
2. Age less than 18 years
3. Inability to provide informed written consent for participation in the study
4. Mean PA less than or equal to 25mmHg or PVR less than 3 wood units
5. PCW greater than 16 mmHg unless increase accounted for by increased transpulmonary gradient greater than or equal to 10 mmHg
6. Patients receiving more than 1 year of oral therapy or more than 6 months of IV therapy.

INCLUSION CRITERIA FOR PATIENTS WITH NONVASCULAR INJURY-INDUCED PULMONARY HYPERTENSION:

The inclusion criteria are as follows:

Patients diagnosed with pulmonary hypertension not known to have histopathology similar to the primary form. Etiologies are listed below.

1. Congenital or acquired valvular or myocardial disease
2. Pulmonary parasitic diseases
3. Arterial hypoxemia with hypercapnea
4. COPD with hypoxemia and forced expiratory volume/forced vital capacity (FEV1/FVC) greater than 2 standard deviations from normal
5. Interstitial lung disease with reduced total lung capacity greater than 2 standard deviations from normal and infiltrates on chest x-ray
6. Pulmonary thromboembolic disease as evidenced by lung perfusion scan or pulmonary angiogram, or intravenous drug abuse
7. Pulmonary hypertension due to congenital abnormalities of the lungs, thorax and diaphragm

EXCLUSION CRITERIA FOR PATIENTS WITH NONVASCULAR INJURY INDUCED PULMONARY HYPERTENSION:

1. Pregnant women (all women of childbearing age will be required to have a screening urine or blood pregnancy test)
2. Age less than 18 years
3. Inability to provide informed written consent for participation in the study
4. Mean PA less than or equal to 25mmHg or PVR less than 3 wood units

EXCLUSION CRITERIA FOR MRI IN SUBJECTS WITH PULMONARY HYPERTENSION:

1) Implanted cardiac pacemaker or defibrillator

2) Central nervous system aneurysm clips

3) Cochlear implants

4) Neural stimulator

5) Ocular foreign body (e.g. metal shavings)

6) Insulin pump

7) Metal shrapnel or bullets

8) Claustrophobia.

Furthermore, the following patient groups will be excluded from studies involving the administration of MRI contrast agents:

1) lactating women

2) renal disease (CrCl less than 20 ml/min)

The creatinine clearance (CrCl) will be calculated using the Cockroft formula where age is in years, kg is weight in kilograms, and Cr is the serum creatinine. If there is no history of kidney disease from the patient or referring physician, additional testing will not be performed. If a patient has a history of renal insufficiency, a recent blood Cr will be used unless the physician performing the test believes the Cr may have changed since the last test. If the Cr may have changed, a blood sample will be obtained for Cr or the subject will be excluded from receiving gadolinium.

CrCl = (140-age) (wt in kg)/72 X serum Cr (mg/dl) for men

CrCl = (0.85) (140-age) (kg)/72 X serum Cr (mg/dl) for women

INCLUSION CRITERIA FOR CONTROL SUBJECTS:

1. Any healthy man or woman who is the appropriate age, race, and gender for matching to a PAH patient
2. No history of HIV infection
3. EKG and echocardiogram with no evidence of clinically relevant heart disease
4. Spirometry with no evidence of clinically relevant lung disease
5. No history of causes of pulmonary hypertension such as collagen vascular disease, chronic liver disease with ALT or AST greater than 2 times the upper limit of normal or cirrhosis of the liver, chronic thromboembolic disease, congenital heart defects, or pulmonary parenchymal disease with hypoxemia
6. No history of diseases thought to be related to development of endothelial dysfunction including systemic hypertension or diabetes requiring drug therapy, hypercholesterolemia and obesity
7. No history of anemia, thrombocytopenia or coagulopathy
8. No history of renal insufficiency
9. No medical conditions requiring chronic medication use with the exception of:

   a. Heartburn, GERD

   b. Environmental allergies, post nasal drip or non-allergic rhinitis

   c. Asthma with no history of oral steroid use, weekly inhaled steroids, or hospitalization for asthma exacerbation

   d. Dermatologic conditions that do not require the use of oral steroids or other immunosuppressants

   e. Treated and stable thyroid disease, depression, or anxiety.
10. No more than 20 cigarettes per years for the previous 2 years and no cigarette use for 30 days prior to the screening evaluation until completion of the study

EXCLUSION CRITERIA FOR CONTROL SUBJECTS:

1. Current pregnancy, lactation or women not currently using medically acceptable birth control. (All women of childbearing age will be required to have a screening urine or blood pregnancy test)
2. Contraindication to MRI scanning including individuals with the following devices:

   A) Implanted cardiac pacemaker or defibrillator

   B) Central nervous system aneurysm clips

   C) Cochlear implants

   D) Implanted Neural stimulator

   E) Ocular foreign body (e.g. metal shavings)

   F) Insulin pump

   G) Metal shrapnel or bullet

   H) Claustophobia
3. Contraindications to MRI contrast agent administration
4. Inability to provide informed written consent for participation in the study
5. Chronic, medically refractory atrial tacharrhythmias
6. Symptoms of heart failure.
7. Mean PA greater than 25mmHG or PVR greater than 1.5 wood units, or PCWP greater than 15 mmHg
8. History of recreational drug use with the exception of marijuana. No marijuana use within 3 months of protocol screening through completion of the study.
9. Intravenous drug abuse.

Volunteers may be excluded if in the opinion of the study investigators they have a condition that may adversely affect the outcome of the study or the safety of the volunteer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-05-17 (Actual); Primary Completion 2009-07-08 (Actual); Study Completion 2009-07-08 (Actual)

PRIMARY OUTCOMES:
Establish the best technique for CEC and PBMC identification, quantification, and isolation and EPC identification and quantification. | one year
  genome-wide expression profiles

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Solomon, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are working on deciding if we want to share IPD.

REFERENCES:
- [Background] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- [Background] International PPH Consortium; Lane KB, Machado RD, Pauciulo MW, Thomson JR, Phillips JA 3rd, Loyd JE, Nichols WC, Trembath RC. Heterozygous germline mutations in BMPR2, encoding a TGF-beta receptor, cause familial primary pulmonary hypertension. Nat Genet. 2000 Sep;26(1):81-4. doi: 10.1038/79226. PMID 10973254
- [Background] Rubin LJ. Primary pulmonary hypertension. Chest. 1993 Jul;104(1):236-50. doi: 10.1378/chest.104.1.236. No abstract available. PMID 8325077
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-CC-0041.html